CLINICAL TRIAL: NCT03716817
Title: Clinical Evaluation of Chairside CAD/CAM Resilient Ceramic Crowns
Brief Title: TetricCAD Crown Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Dennis J. Fasbinder, DDS, Clinica Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00145596
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Fractured Tooth; Decayed Tooth; Unsatisfactory Restoration of Tooth
Keywords: Crown; Ceramic; CAD/CAM
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tetric CAD Crown (Experimental): Tetri CAD crowns will hand polished and cemented with a dual cured resin cement (Variolink Esthetic by Ivoclar Vivadent).
  Interventions: Device: Tetric CAD

INTERVENTIONS:
Device: Tetric CAD — Resilient ceramic crowns (Tetric CAD by Ivoclar Vivadent) are placed using an adhesive bonding process including a total etch process with a universal adhesive (Adhese by Ivoclar Vivadent) and dual cured resin cement (Variolink Esthetic by Ivoclar Vivadent).

SUMMARY:
This investigation will be a clinical trial to study the performance of a new resin-based ceramic material for crowns. The material has been approved by the FDA for patient treatment. A computer technique will be used to fabricate the crowns in a single appointment without the need for a temporary crown or second appointment. The purpose of the study is to measure how well the high strength crowns function over an extended period of time.

DETAILED DESCRIPTION:
The study will be composed of 50 crowns placed in adult patients that have been identified as requiring at least one crown on a posterior tooth. A maximum of two crowns per patient will be completed. All the crowns will be made from the same resilient ceramic CAD/CAM block(Tetric CAD/Ivoclar Vivadent). The crowns are placed using an adhesive bonding process including a total etch process with a universal adhesive (Adhese by Ivoclar Vivadent) and dual-cured resin cement (Variolink Esthetic by Ivoclar Vivadent). The crowns are planned to be evaluated at 6 months, 1 year, 2 years, 3 years, and if funding permits, 4 years, and 5 years. At each appointment, an examination of the crown will be completed as well as clinical photographs, an intraoral digital scan, and impression of the crown.

ELIGIBILITY:
Inclusion Criteria:

* must have at least one carious lesion or defective restoration or fractured tooth in a molar or premolar
* reason for restoration should extend more than one-half the intercuspal width of the tooth requiring a full crown restoration
* Teeth to be vital and asymptomatic prior to treatment
* No more than two restorations will be placed per patient. If a patient presents with more than two acceptable teeth for the study, molar teeth will be included prior to premolar teeth.

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth with prior endodontic treatment of any kind
* Teeth with a history of direct or indirect pulp capping procedures
* Patients with significant untreated dental disease to include periodontitis and rampant caries
* Pregnant or lactating women
* Patients with a history of allergies to any of the materials to be used in the study
* Patients unable to return for the recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Crown failure | from delivery of the crown up to 5 years
  Crown failure includes fracture of the crown or loss of the crown requiring placement of a new crown at any time between delivery and five years.

SECONDARY OUTCOMES:
Crown loss of retention | from delivery of the crown up to 5 years
  Loss of retention is measured as detachment of the crown from the tooth without fracture of the crown requiring recementation of the crown.
Tooth sensitivity | from delivery of the crown up to 5 years
  Patient described sensitivity on a scale of 1 to 4, where 1 means absence of sensitivity (pain) and four means severe discomfort noted routinely with cold or pressure stimulation.
Margin staining | from delivery of the crown up to 5 years
  Margin staining is categorized based on modified US Public Health Service criteria using a four point scale where 1 is no staining and 4 is penetrating stain involving more than 50% of the margin.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No